CLINICAL TRIAL: NCT06877507
Title: Rapid Diagnostic Technology for Acute Upper Gastrointestinal Bleeding Based on Analysis of Volatile Organic Compounds (VOCs) in Exhaled Breath
Brief Title: Rapid Diagnostic Technology for AUGIB Based on Analysis of VOCs in Exhaled Breath
Acronym: VOCsAUGIB
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 302-2025-VOCs; 82270694 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Volatile Organic Compound; Gastrointestinal Hemorrhage
Keywords: Volatile Organic Compound; Acute Upper Gastrointestinal Bleeding; Exhaled Breath
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — exhaled breath
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- No bleeding: No blood in the upper gastrointestinal tract
  Interventions: Device: Gastroscopy; Diagnostic Test: Gas Chromatography - Mass Spectrometry
- Minor bleeding: A little blood in the upper gastrointestinal tract
  Interventions: Device: Gastroscopy; Diagnostic Test: Gas Chromatography - Mass Spectrometry
- Major bleeding: Plenty of blood in the upper gastrointestinal tract
  Interventions: Device: Gastroscopy; Diagnostic Test: Gas Chromatography - Mass Spectrometry

INTERVENTIONS:
Device: Gastroscopy — Gastroscopy for all included patients
Diagnostic Test: Gas Chromatography - Mass Spectrometry — Using a patient's exhaled breath test with Gas Chromatography - Mass Spectrometry

SUMMARY:
This study aims to develop a non-invasive and rapid diagnostic technology for acute upper gastrointestinal bleeding (AUGIB) by analyzing volatile organic compounds (VOCs) in exhaled breath. Clinically confirmed patients will be divided into three groups (no bleeding, minor bleeding, major bleeding) based on endoscopic findings. VOC profiles will be analyzed to construct a predictive model, validated for sensitivity and specificity (both targets ≥0.7). This approach addresses the limitations of endoscopy in emergency or resource-limited settings, improving diagnostic efficiency and reducing mortality.

DETAILED DESCRIPTION:
Acute upper gastrointestinal bleeding (AUGIB) is a common emergency with an annual incidence of 100-180/100,000 and mortality of 2%-15%. Endoscopy, the gold standard, is invasive and equipment-dependent, limiting its use in primary care or emergencies. Exhaled breath VOCs analysis, a non-invasive and portable method, has been applied in other diseases but not yet explored for AUGIB.

Objectives:

1. Identify characteristic VOC profiles in exhaled breath of AUGIB patients.
2. Develop a VOC-based predictive model with sensitivity and specificity ≥0.7.
3. Establish rapid diagnostic criteria to enhance clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Clinical suspicion of AUGIB (e.g., hematemesis, melena);
3. Fasting ≥4 hours;
4. Signed informed consent.

Exclusion Criteria:

1. Severe pulmonary dysfunction or recent lung infection (within 1 week);
2. Cardiac/renal failure or disseminated intravascular coagulation;
3. Contraindications to endoscopy;
4. High-risk conditions (e.g., massive ascites);
5. Alcohol consumption within 24 hours;
6. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring endoscopy for suspected AUGIB
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the diagnostic model | 4 months
  targets ≥0.7

SECONDARY OUTCOMES:
Identification of key VOCs | 4 months
  e.g., aldehydes, ketones
Differences in VOC concentrations across 3 bleeding severity groups | 4 months
  Different VOCs